CLINICAL TRIAL: NCT03097835
Title: Evaluation of Skin Quality Improvement When Hyper-Diluted OnabotulinumtoxinA (Botox®, Botox® Cosmetic /BTXa/) is Injected Into The Superficial Dermis of the Mid-Face
Brief Title: Evaluation of Skin Quality Improvement
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Steve Yoelin M.D. Medical Associates, Inc. (Other)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HDB101
Record Dates: First submitted 2017-03-27; First posted 2017-03-31 (Actual); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Skin Quality
MeSH Terms: interventions — Anesthesia; Saline Solution

STUDY DESIGN:
Intervention Model Description: This will be a longitudinal study in which patients will be initially treated with hyper-diluted Botox Cosmetic in the superficial dermis or they will be treated 0.9% saline. Then, on day 30 of the study patients initially treated with hyper diluted Botox Cosmetic will be treated with saline and patients initially treated with saline will be treated with hyper-diluted botox.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A (Other): Group A will be treated with Hyper-Diluted Botox on day 1 and on day 30 they will be treated with 0.9% saline solution.
  Interventions: Drug: Hyper-Diluted Botox; Drug: Topical anesthesia; Other: 0.9% saline solution
- Group B (Other): Group B will be treated with 0.9% saline solution on day 1 and on day 30 they will be treated with Hyper-Diluted Botox.
  Interventions: Drug: Hyper-Diluted Botox; Drug: Topical anesthesia; Other: 0.9% saline solution

INTERVENTIONS:
Drug: Hyper-Diluted Botox — 0.1ml of hyper-diluted Botox® Cosmetic will be administered in the superficial dermis using a 1ml luer lock syringe coupled with a 33g ½" needle
Drug: Topical anesthesia — Topical anesthesia will be bilaterally applied to the mid-face region for 20 minutes
Other: 0.9% saline solution — 0.1ml of 0.9% saline solution will be administered to the side of the face

SUMMARY:
The purpose of this study is to comprehensively investigate and objectively demonstrate the effectiveness of hyperdiltue Botox® Cosmetic in improving overall skin quality, more specifically evenness of skin tone, reduction of pore size and improvement in the appearance of preexisting skin scars.

DETAILED DESCRIPTION:
The purpose of this study is to comprehensively investigate and objectively demonstrate the effectiveness of hyperdiltue Botox® Cosmetic in improving overall skin quality, more specifically evenness of skin tone, reduction of pore size and improvement in the appearance of preexisting skin scars. The ability of hyperdilute Botox® Cosmetic to improve overall skin quality is likely optimized when it is injected uniformly in hyper-diluted small aliquots in order to "saturate" the dermis. We propose to prepare Botox® Cosmetic in a manner that is approximately 4 times more dilute compared to the typical Botox® Cosmetic preparation. A 4x4 centimeter area located in the mid-cheek adjacent to the nose will be injected with hyperdilute Botox® Cosmetic. Botox® Cosmetic is not FDA-approved for this use. A maximum of 15 subjects will participate in this study, all of whom will receive injections of Botox® Cosmetic during the course of this study.

This study is a randomized, placebo-controlled, and double-masked study. This means neither the study doctor nor participant know the experimental agent (e.g., 0.9% saline solution and hyperdiluted Botox® Cosmetic) injected on each side of the patients' faces. The study will last for a total of 75 days. Evaluation of the study is based on the analysis of photographic images obtained during the study.

ELIGIBILITY:
Inclusion Criteria:

* Ability to follow study instructions and likely to complete all required visits
* Written consent has been obtained
* Written authorization for "Use and Release of Health and Research Study Information" has been obtained
* Subjects who are Fitzpatrick Skin Types II-IV

Exclusion Criteria:

* Subjects must be Onabotulinum Toxin Type A naive; if subject has had Onabotulinum Toxin Type A administered in the face in the previous 12 months they are excluded
* Subjects must be dermal filler naïve in the lateral canthal region and midface regions
* Subjects must be energy or light device naïve
* Subjects must have average or below-average lifetime sun exposure
* Subjects must be free of inflammatory skin disease(s)

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Females of reproductive age must use acceptable and reliable forms of birth control Females of reproductive age must undergo urine pregnancy testing
Enrollment: 15 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2018-07-12 (Actual); Study Completion 2018-07-26 (Actual)

PRIMARY OUTCOMES:
Percent Improvement in Skin Quality | Entire duration of the study (Day 1-Day 135)
  An evaluation of the percent improvement in skin quality when the "Onabotulinum Toxin Type A" treated side of face is compared to the "placebo" treated side of the face. Good skin quality is defined as small pore size, evenness of skin texture, evenness of skin tone, minimal presence of wrinkles, and minimal presence of scars. We will measure improvement primarily by image analysis of the photos taken during each visit using the Canfield Scientific camera (or the Allergan provided alternative).

SECONDARY OUTCOMES:
Patient and Investigator Reported Outcomes | Entire duration of the study (Day 1-Day 135)
  An objective observer as well as the patient will evaluate if there is an improvement in skin quality throughout the course of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Steve Yoelin MD & Associates, Newport Beach, California, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared through the form of either a published paper or poster presentation.

REFERENCES:
- [Result] Bansal C, Omlin KJ, Hayes CM, Rohrer TE. Novel cutaneous uses for botulinum toxin type A. J Cosmet Dermatol. 2006 Sep;5(3):268-72. doi: 10.1111/j.1473-2165.2006.00255.x. PMID 17177750
- [Result] Diamond A, Jankovic J. Botulinum toxin in dermatology - beyond wrinkles and sweat. J Cosmet Dermatol. 2006 Jun;5(2):169. doi: 10.1111/j.1473-2165.2006.00250.x. No abstract available. PMID 17173593
- [Result] Xiao Z, Zhang F, Lin W, Zhang M, Liu Y. Effect of botulinum toxin type A on transforming growth factor beta1 in fibroblasts derived from hypertrophic scar: a preliminary report. Aesthetic Plast Surg. 2010 Aug;34(4):424-7. doi: 10.1007/s00266-009-9423-z. Epub 2009 Oct 3. PMID 19802513